CLINICAL TRIAL: NCT05985668
Title: Towards Improved Diagnostics for Suspected Platelet Function Disorders
Status: Recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: K-2023-0991
Record Dates: First submitted 2023-06-30; First posted 2023-08-14 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-06

CONDITIONS: Platelet Function Disorder; Platelet Disorder; Thrombocytopathy
Keywords: diagnostic accuracy
MeSH Terms: conditions — Blood Platelet Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Suspected: Suspected Platelet Function Disorder during bleeding investigation
- Confirmed: Confirmed Platelet Function Disorder by Functional or Genetic Assay, or confirmed negative by gold standard assay

SUMMARY:
This study aims to improve platelet function testing during bleeding investigations. To this end, the study will evaluate the diagnostic accuracy of novel platelet function tests in patients with confirmed or suspected platelet function disorders. Study participants will be recruited from patients that are referred to or treated at the Coagulation Unit, Karolinska University Hospital, and Pediatric Coagulation Unit, Astrid Lingren Children's Hospital.

ELIGIBILITY:
Inclusion Criteria, known defects:

* Known platelet function disorder under follow-up at Karolinska University Hospital (genetic or functional assay)
* High likelihood of platelet function disorder (aberrant screening test with inheritance)
* Family investigation for platelet disorder

Exclusion Criteria, known defects::

* Antiplatelet or anticoagulant drugs
* vWF:GPIb below 0.40 IU/mL
* Hematocrit below 0.35 or above 0.50
* Other coagulation disorder

Inclusion Criteria, suspected platelet function disorder:

* Bleeding investigation at Karolinska University Hospital

Exclusion Criteria, suspected platelet function disorder::

* Antiplatelet or anticoagulant drugs
* vWF:GPIb below 0.40 IU/mL
* Hematocrit below 0.35 or above 0.50
* Other coagulation disorder

Min Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients recruited at Karolinska University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Platelet-thrombus formation on collagen surface | At study inclusion
  Whole-blood platelet-thrombus formation on collagen surface measured in a semi-automatic microchip flow chamber by a pressure sensor. Coagulation activation is inhibited.

OTHER OUTCOMES:
Platelet count effect on platelet-thrombus formation on collagen surface | At study inclusion
  Whole-blood platelet-thrombus formation on collagen surface as for primary outcome. Subgroup analysis for patients with platelet count < 150 x 10^9 /L.
ddAVP effect on platelet-thrombus formation on collagen surface | Immediately before and 1 hour after administration of ddAVP.
  Whole-blood platelet-thrombus formation on collagen surface, similar as for primary outcome measurement. In a subset of patients with a clinical indication (physician discretion).
Thrombus formation on collagen/TF | At study inclusion
  Thrombus formation on collagen surface/tissue-factor surface measured in a semi-automatic microchip flow chamber by a pressure sensor.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes